CLINICAL TRIAL: NCT00524979
Title: Digital Voice Analysis in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: Ilana Vaintrayb, MD, BeerYaakov Mental Health Center
Other Study IDs: Voice -200CTIL
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Schizophrenia: People who are diagnosed as schizophrenic by DSM-IV
- Mental diseases: Patients who are deagnosed as having mental disease other then schizophrenia
- Mentally healthy: People who have no mental disease

SUMMARY:
There is a differences in voice frequency of schizophrenic patients compared to patients with other mental diseases and compared to mentally healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic patients
* Other mental disease patients
* Healthy people
* People above age 18

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Schizophrenic patients
  * Other mental disease patients
  * Healthy people
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-10; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Vaintraub, MD, Principal Investigator — Beer Yaakov Mental Health Center
Locations (1):
- Beer Yaakov MHC, Beer Yaakov, Beer Yaakov, Israel